CLINICAL TRIAL: NCT04113720
Title: The Effects of Levobupivacaine Versus Levobupivacaine Plus Dexmedetomidine Infiltration for Post-tonsillectomy Analgesia and Laryngospasm in Pediatric Patients
Brief Title: Levobupivacaine vs Levobupivacaine + Dexmedetomidine Infiltration for Post-tonsillectomy Analgesia and Laryngospasm in Pediatric Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300316
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Post-tonsillectomy Analgesia; Levobupivacaine
MeSH Terms: interventions — Levobupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): children will receive levobupivacaine 0.25% by peritonsillar infiltration after intubation 3- 5 min before the start of surgery.
  Interventions: Drug: Levobupivacaine hydrochloride
- Group B (Active Comparator): children will receive levobupivacaine 0.25% plus dexmedetomidine 1µg/kg diluted in 4 ml saline 0.9% and given by peritonsillar infiltration (2 ml per tonsil), after intubation 3- 5 min before the start of surgery.
  Interventions: Drug: Levobupivacaine Hydrochloride + Dexmedetomidine

INTERVENTIONS:
Drug: Levobupivacaine hydrochloride — levobupivacaine 0.25%
  Other Names: levobupivacaine
  Arms: Group A
Drug: Levobupivacaine Hydrochloride + Dexmedetomidine — Levobupivacaine plus Dexmedetomidine
  Other Names: levobupivacaine + precedex
  Arms: Group B

SUMMARY:
Tonsillectomy is one of the most common surgical performed procedures in children. Adenotonsillectomy surgery in pediatrics is commonly managed as an ambulatory surgery. This may be attributed to the use of the electro-dissection surgical technique that decreases the incidence of immediate postoperative hemorrhage. However, the use of the electro-cautery technique increases postoperative inflammation. Postoperative throat pain is a very important and significant problem because it can lead to decreased oral intake and dehydration with subsequent serious complications of dehydration.

DETAILED DESCRIPTION:
The idea behind the use of local anesthetic agents in the peri-operative period is not only related to its ability to block peripheral nociceptor transmission after tissue damage but also in preventing sensitization of the central nervous system. Levobupivacaine is new, long-acting bupivacaine, amide-type local anesthetic and is thought to be less cardio and neurotoxic. However, few studies showed that local infiltration of levobupivacaine reduces the intensity of postoperative pain. Dexmedetomidine is a highly selective α2-adrenoceptor agonist recently introduced to anesthesia practice producing dose-dependent sedation, anxiolysis, and analgesia (involving spinal and supraspinal sites), without respiratory depression. Dexmedetomidine is being used off-label as an adjunctive agent in pediatric patients for sedation and analgesia; in the critical care unit, during non-invasive ( Magnetic resonance imaging) and invasive procedures ( cardiac catheterization and endoscopy). It may also decrease opioid usage and anesthesia requirements as seen from adult data prevent emergence delirium and postanesthesia shivering.

ELIGIBILITY:
Inclusion Criteria:

* Weight: 10-40 kg
* American Society of Anesthesiologists ASA physical status: I-II.
* Operation: elective tonsillectomy (±adenoidectomy) in the otorhinolaryngology department, Assuit University Hospitals due to recurrent or chronic tonsillitis with or without adenoidectomy (using the surgical retraction and bipolar diathermy if indicated).

Exclusion Criteria:

* Patients having known hypersensitivity to dexmedetomidine or levobupivacaine.
* Patients with the following conditions: obstructive sleep apnea syndrome (whether confirmed by a polysomnography test or not), previous peritonsillar abscess formation and those with swallowing disorders.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
the first call for rescue analgesia | in 24 hours.
  pain assessment using the CHEOPS scale

SECONDARY OUTCOMES:
The analgesics consumption | in 24 hours.
  The total analgesics consumption
parental satisfaction | 24 hours
  a five-point Likert scale (1 - very dissatisfied, 2 - dissatisfied, 3 - neutral, 4 - satisfied, 5 - very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akoglu E, Akkurt BC, Inanoglu K, Okuyucu S, Dagli S. Ropivacaine compared to bupivacaine for post-tonsillectomy pain relief in children: a randomized controlled study. Int J Pediatr Otorhinolaryngol. 2006 Jul;70(7):1169-73. doi: 10.1016/j.ijporl.2005.12.001. Epub 2006 Jan 18. PMID 16414124
- [Background] Arbin L, Enlund M, Knutsson J. Post-tonsillectomy pain after using bipolar diathermy scissors or the harmonic scalpel: a randomised blinded study. Eur Arch Otorhinolaryngol. 2017 May;274(5):2281-2285. doi: 10.1007/s00405-017-4451-9. Epub 2017 Feb 17. PMID 28213775
- [Background] Blaine Easley R, Brady KM, Tobias JD. Dexmedetomidine for the treatment of postanesthesia shivering in children. Paediatr Anaesth. 2007 Apr;17(4):341-6. doi: 10.1111/j.1460-9592.2006.02100.x. PMID 17359402
- [Background] Karaaslan K, Yilmaz F, Gulcu N, Sarpkaya A, Colak C, Kocoglu H. The effects of levobupivacaine versus levobupivacaine plus magnesium infiltration on postoperative analgesia and laryngospasm in pediatric tonsillectomy patients. Int J Pediatr Otorhinolaryngol. 2008 May;72(5):675-81. doi: 10.1016/j.ijporl.2008.01.029. Epub 2008 Mar 5. PMID 18325601